CLINICAL TRIAL: NCT03981900
Title: IDentification of Predictive Factors of Continuation of Treatment With Tofacitinib in Patients With Rheumatoid Arthritis in Common Practice and the Impact of the Patient's Behavioural Strategies on Clinical Parameters: The DeFacTo Study.
Brief Title: IDentification of Factors Predictive of Tofacitinib's Survival in Patient With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921313; DeFacTo (Other: Alias Study Number)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis: All participants with a diagnosis of moderate to severe active rheumatoid arthritis and treated with Tofacitinib
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — 5 mg BID, oral administrtaion
  Other Names: Xeljanz
Drug: Tofacitinib — tablet form 11mg once daily oral
  Other Names: Xeljanz

SUMMARY:
Regarding Tofacitinib, newly introduced on the market, few data on drug retention and no data on the factors predictive of Tofacitinib drug survival in patients with RA are available.

Therefore, the primary objective of the DeFacTo study will be to identify the factors predictive of Tofacitinib drug survival in patients with RA.

As secondary objectives, the impact of behavioural strategies on drug survival and other clinical parameters as well as Tofacitinib effectiveness and tolerability will be studied under real-life conditions of use in French patients with RA.

DETAILED DESCRIPTION:
This is an observational, open-label, prospective, multi-centre, national study designed to evaluate the factors predictive of Tofacitinib's survival in patients with rheumatoid arthritis

If catastrophisation is described as a distortion of the perception of pain involving a both emotional and cognitive component, pushing the patient to see only the worst, coping involves adaptive strategies by which the patient attempts to find solutions in order to better cope with his/her disease. It has been demonstrated that such behavioural strategies can influence directly or indirectly the intensity of symptoms in patients suffering from chronic disease.

Therefore, as secondary objectives, the impact of behavioural strategies on drug survival and other clinical parameters as well as Tofacitinib effectiveness and tolerability will be studied under real-life conditions of use in French patients with RA.

The duration of this study will be approximately 48 months including a 24-month recruitment period and a 24-month patient follow-up period.

Patients will be followed prospectively and follow-up visits will be conducted after the initial consultations. No visit or additional test is required by the protocol, since the study is observational

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient in whom the diagnosis of moderate to severe active rheumatoid arthritis has been confirmed by a rheumatologist
* Patient for whom the rheumatologist decides to initiate treatment with Tofacitinib
* Patient informed of the study

Exclusion Criteria:

* Patient participating in a randomised clinical trial.
* Patient presenting with a contraindication to prescription of Tofacitinib
* Patients who are investigational site staff members or patients who are Pfizer employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of moderate to severe active rheumatoid arthritis for whom the rheumatologist has decided to initiate a treatment with Tofacitinib
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (66):
- France (66):
  - Centre Hospitalier D'arras, Arras
  - Hopital Robert Ballanger, Aulnay-sous-Bois
  - Cabinet Medical, Aurillac
  - Centre Hospitalier D Auxerre, Auxerre
  - Institut Calot Helio Marin, Berck
  - hopital Avicenne, Bobigny
  - Centre Hospitalier de Fleyriat, Bourg-en-Bresse
  - Hopital Jacques Cœur, Bourges
  - Cabinet Medical, Brest
  - Cabinet Medical, Brive-la-Gaillarde
  - Cabinet Medical, Bruges
  - Centre Hospitalier Jean Rougier, Cahors
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Hopital Pierre Nouveau, Cannes
  - Centre Hospitalier de Carcassonne, Carcassonne
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier de Compiegne, Compiègne
  - Hopital Henri Mondor, Créteil
  - Hopital Victor Jousselin, Dreux
  - Centre Hospitalier des Deux Vallees Juvisy, Juvisy-sur-Orge
  - Cabinet Medical, La Battie Vieille
  - Cabinet Medical, La Moutonne
  - Centre Hospitalier Departemental Vendee Les Oudairies, La Roche-sur-Yon
  - Hopital Suburbain Du Bouscat, Le Bouscat
  - Hopital Suburbain, Le Bouscat
  - Centre Hospitalier Universitaire de Lille - Hopital B Roger Salengro, Lille
  - Hopital B Roger Salengro-chu De Lille, Lille
  - Hopital Dupuytren, Limoges
  - Cabinet Medical, Limoges
  - Clinique de La Sauvegarde / Cabinet Le Trait D Union, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Clinique du Pont de Chaume, Montauban
  - Centre Hospitalier de Montauban, Montauban
  - Centre Hospitalier Montceau Les Mines-Hopital Jean Bouveri, Montceau-les-Mines
  - Hopital Jacques Monod, Montivilliers
  - Cabinet Medical, Montpellier
  - Cabinet Medical Saint Roch, Montpellier
  - Clinique Beau Soleil, Montpellier
  - Hopital Lapeyronie, Montpellier
  - Hopital Caremeau, Nîmes
  - Centre Hospitalier Orleans-Hopital La Source, Orléans
  - Cabinet Medical, Paris
  - Centre Hospitalier Pitie Salpetriere, Paris
  - Hopital Cochin, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Centre Hospitalier de Perigueux, Périgueux
  - Hospices Civils de Lyon - Hopital Lyon Sud- Hematologie, Pierre-Bénite
  - Cabinet Medical, Poitiers
  - Centre Hospitalier La Miletrie, Poitiers
  - Centre Hospitalier Annecy Genevois Site Annecy, Pringy
  - Hopital Charles Nicolle, Rouen
  - Cabinet Medical, Saint-Lô
  - Hopital Inter-armees Begin, Saint-Mandé
  - Centre Hospitalier Universitaire Saint Pierre, Saint-Pierre
  - Centre Hospitalier Universitaire Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Nord, Saint-Priest-en-Jarez
  - Centre Hospitalier de Bigorre Site La Gespe, Tarbes
  - Clinique Medipole Garonne, Toulouse
  - Hopital Purpan, Toulouse
  - Cabinet Medical, Toulouse
  - Cabinet de Rhumatologie, Tours
  - Cabinet Medical, Tours
  - Hopital des Hauts Clos, Troyes
  - Cabinet Medical, Valenciennes
  - Hopital Psv, Villeneuve-sur-Lot
  - Cabinet Medical, Vincennes

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with moderate-to-severe active rheumatoid arthritis who initiated Tofacitinib in the real-world setting were observed in this study.
Groups:
- Tofacitinib: Participants with rheumatoid arthritis who received tofacitinib were included in this observational study. The recommended dosage is one Tofacitinib 5 milligram (mg) tablet (immediate release tablets) twice daily or Tofacitinib 11 mg (extended-release tablets) once a day, the transition from one formulation to another is possible according to the recommendations mentioned in the summary of product characteristics (SmPC).
Period: Overall Study
Arm/Group | Tofacitinib
Started | 314
Safety Analysis Set (SAS) | 309
Full Analysis Set (FAS) | 306
Completed | 227
Not Completed | 87
Not completed — Participant decision - Without withdrawal of consent | 17
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 46
Not completed — Decision of the researcher | 3
Not completed — Death | 3
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included participants who received at least one dose of Tofacitinib.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 309
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 194
  >= 65 Years | 112
  Missing | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 241
  Male | 65
  Missing | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Duration of Tofacitinib Drug Survival
Description: The duration of tofacitinib drug survival was calculated as: date of permanent drug discontinuation minus date of first taking the drug + 1. If a participant did not present with the event of interest, that is they did not have a permanent drug discontinuation record during the study, then they were censored at the time of their last visit. Kaplan-Meier method was used for estimation.
Time Frame: Date of initiation of study drug treatment up to date of permanent drug discontinuation or date of censoring (up to a maximum of 48 months)
Population: Full analysis set population included participants who met the eligibility criteria, received at least one dose of Tofacitinib and had at least one set of post-baseline measurements.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Months | 26.4 [24.1 to NA] — Data for the upper limit of 95% CI was not estimable due to insufficient follow-up in this study.

2. Secondary Outcome: Change From Baseline in Total Pain Catastrophising Scale (PCS) Score at Month 1, 3, 6, 12, 18 and 24
Description: PCS is a 13 item questionnaire around thoughts and emotions experienced during pain, with each question scored on a 5-point scale ranging from 0 (not at all) to 4 (all the time), where higher scores indicated worse condition. There are three subscales of PCS: rumination (thinking deeply) [4 items], exaggeration [3 items] and helplessness [6 items]. Total scores and domain scores are derived by summing the scores of the individual items. Overall possible Total PCS score range is 0 to 52, where higher scores signifies worse condition. A total score of greater than or equal to (>=) 20 indicates a clinically relevant level of catastrophising. Mean change from baseline in total PCS score is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18 and 24
Population: Full analysis set population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. Here, "Number of participants analyzed" signifies number of participants evaluable and contributed to data for this outcome measure. Here, "Number Analyzed" signifies number of participants evaluable at specified time points. No imputation used for missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 231
Units on a scale
  Baseline | 20.4 (14.0)
  Change at Month 1: number analyzed (Participants) | 152
  Change at Month 1 | -5.2 (10.4)
  Change at Month 3: number analyzed (Participants) | 161
  Change at Month 3 | -6.6 (11.1)
  Change at Month 6: number analyzed (Participants) | 137
  Change at Month 6 | -8.4 (11.4)
  Change at Month 12: number analyzed (Participants) | 110
  Change at Month 12 | -8.2 (11.6)
  Change at Month 18: number analyzed (Participants) | 105
  Change at Month 18 | -8.8 (11.2)
  Change at Month 24: number analyzed (Participants) | 91
  Change at Month 24 | -8.7 (10.8)

3. Secondary Outcome: Change From Baseline in Coping Strategies Questionnaire (CSQ) Score at Month 1, 3, 6, 12, 18 and 24
Description: CSQ evaluates cognitive coping, has 21 items and 5 domains in its French version. For each item, participants rate the frequency of their use of each coping strategy on a 4- point Likert-type scale (0= Never, 1= sometimes, 2= often and 3= very often). Domain scores are derived by summing the individual items scores that make-up the domain. Five domains with score range: distraction (5 items, score range: 0 to 15), catastrophising (4 items, score range: 0 to 12), distancing from pain (4 items, score range: 0 to 12), ignoring pain sensations (5 items, score range: 0 to 15) and praying (3 items, score range: 0 to 9). For each domain, higher scores indicated worse condition. Mean change from baseline in CSQ domain scores are reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6 12, 18 and 24
Population: Full analysis set population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. Here, "Number Analyzed" signifies number of participants evaluable at specified time points. No imputation used for missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Units on a scale
  Distraction at baseline: number analyzed (Participants) | 251
  Distraction at baseline | 13.2 (3.8)
  Catastrophising at baseline: number analyzed (Participants) | 247
  Catastrophising at baseline | 8.4 (3.0)
  Distancing from Pain at baseline: number analyzed (Participants) | 246
  Distancing from Pain at baseline | 7.3 (3.2)
  Ignoring Pain Sensations at baseline: number analyzed (Participants) | 247
  Ignoring Pain Sensations at baseline | 11.3 (3.6)
  Praying at baseline: number analyzed (Participants) | 244
  Praying at baseline | 5.6 (2.9)
  Distraction, Change at month 1: number analyzed (Participants) | 170
  Distraction, Change at month 1 | -0.4 (3.3)
  Catastrophising, Change at month 1: number analyzed (Participants) | 168
  Catastrophising, Change at month 1 | -0.6 (2.8)
  Distancing from Pain, Change at month 1: number analyzed (Participants) | 171
  Distancing from Pain, Change at month 1 | -0.0 (2.9)
  Ignoring Pain Sensations, Change at month 1: number analyzed (Participants) | 170
  Ignoring Pain Sensations, Change at month 1 | -0.7 (3.7)
  Praying, Change at month 1: number analyzed (Participants) | 168
  Praying, Change at month 1 | -0.1 (2.2)
  Distraction, Change at month 3: number analyzed (Participants) | 194
  Distraction, Change at month 3 | -0.9 (4.5)
  Catastrophising, Change at month 3: number analyzed (Participants) | 192
  Catastrophising, Change at month 3 | -1.0 (3.3)
  Distancing from Pain, Change at month 3: number analyzed (Participants) | 189
  Distancing from Pain, Change at month 3 | -0.2 (3.9)
  Ignoring Pain Sensations, Change at month 3: number analyzed (Participants) | 187
  Ignoring Pain Sensations, Change at month 3 | -0.2 (4.1)
  Praying, Change at month 3: number analyzed (Participants) | 184
  Praying, Change at month 3 | -0.5 (2.0)
  Distraction, Change at month 6: number analyzed (Participants) | 167
  Distraction, Change at month 6 | -1.5 (4.2)
  Catastrophising, Change at month 6: number analyzed (Participants) | 162
  Catastrophising, Change at month 6 | -1.5 (2.6)
  Distancing from Pain, Change at month 6: number analyzed (Participants) | 163
  Distancing from Pain, Change at month 6 | -0.5 (4.1)
  Ignoring Pain Sensations, Change at month 6: number analyzed (Participants) | 166
  Ignoring Pain Sensations, Change at month 6 | -0.3 (4.4)
  Praying, Change at month 6: number analyzed (Participants) | 163
  Praying, Change at month 6 | -0.7 (2.1)
  Distraction, Change at month 12: number analyzed (Participants) | 134
  Distraction, Change at month 12 | -1.5 (4.3)
  Catastrophising, Change at month 12: number analyzed (Participants) | 133
  Catastrophising, Change at month 12 | -1.8 (2.4)
  Distancing from Pain, Change at month 12: number analyzed (Participants) | 135
  Distancing from Pain, Change at month 12 | -0.6 (3.9)
  Ignoring Pain Sensations, Change at month 12: number analyzed (Participants) | 133
  Ignoring Pain Sensations, Change at month 12 | -0.9 (4.5)
  Praying, Change at month 12: number analyzed (Participants) | 101
  Praying, Change at month 12 | -0.7 (2.2)
  Distraction, Change at month 18: number analyzed (Participants) | 106
  Distraction, Change at month 18 | -1.5 (4.5)
  Catastrophising, Change at month 18: number analyzed (Participants) | 107
  Catastrophising, Change at month 18 | -1.6 (2.7)
  Distancing from Pain, Change at month 18: number analyzed (Participants) | 107
  Distancing from Pain, Change at month 18 | -0.5 (3.3)
  Ignoring Pain Sensations, Change at month 18: number analyzed (Participants) | 107
  Ignoring Pain Sensations, Change at month 18 | -0.8 (4.4)
  Praying, Change at month 18: number analyzed (Participants) | 105
  Praying, Change at month 18 | -0.6 (2.2)
  Distraction, Change at month 24: number analyzed (Participants) | 102
  Distraction, Change at month 24 | -1.6 (5.4)
  Catastrophising, Change at month 24: number analyzed (Participants) | 103
  Catastrophising, Change at month 24 | -1.6 (2.6)
  Distancing from Pain, Change at month 24: number analyzed (Participants) | 100
  Distancing from Pain, Change at month 24 | -0.7 (2.8)
  Ignoring Pain Sensations, Change at month 24: number analyzed (Participants) | 102
  Ignoring Pain Sensations, Change at month 24 | -0.5 (4.4)
  Praying, Change at month 24: number analyzed (Participants) | 101
  Praying, Change at month 24 | -0.7 (2.2)

4. Secondary Outcome: Percentage of Participants With Low Disease Activity (LDA) According to Disease Activity Index 28 (DAS28)-4 Erythrocyte Sedimentation Rate (ESR) (<=3.2)
Description: DAS28-4 ESR is a composite endpoint, calculated using 4 variables (represented by '4' in the name). Components includes: Tender Joint Count (TJC) with 28 joints assessed, Swollen Joint Count (SJC) with 28 joints assessed, ESR (millimeter per hours [mm/h]) and Patient Global Assessment (PtGA) recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). The calculation of DAS28-4 ESR is as follows: 0.56 * square root (sqrt) (TJC) + 0.28 * sqrt (SJC) + 0.70* In (ESR) + 0.014* (PtGA); where ln = natural logarithm. Total DAS28-4 score range: 0 to 9.4, higher score=more disease activity. DAS28(ESR) score of <=3.2 indicates LDA. Percentage of participants with DAS28-4 ESR <=3.2 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 249
  Baseline | 7.2
  Month 1: number analyzed (Participants) | 152
  Month 1 | 34.9
  Month 3: number analyzed (Participants) | 196
  Month 3 | 46.4
  Month 6: number analyzed (Participants) | 166
  Month 6 | 52.4
  Month 12: number analyzed (Participants) | 135
  Month 12 | 57.0
  Month 18: number analyzed (Participants) | 116
  Month 18 | 55.2
  Month 24: number analyzed (Participants) | 103
  Month 24 | 60.2

5. Secondary Outcome: Percentage of Participants With LDA According to DAS28-4 C Reactive Protein (CRP) (<=3.2)
Description: DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC with 28 joints assessed, SJC with 28 joints assessed, CRP (mg/L) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). The calculation of DAS28-4 CRP is as follows: 0.56 * sqrt (TJC) + 0.28 * sqrt (SJC) + 0.36 * ln (CRP+l) + 0.014*PtGA + 0.96; where ln = natural logarithm. Total DAS28-4 score range: 0 to 9.4, higher score=more disease activity. DAS28(CRP) score of <=3.2 indicates LDA. Percentage of participants with DAS28-4 CRP <=3.2 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 286
  Baseline | 9.8
  Month 1: number analyzed (Participants) | 184
  Month 1 | 46.2
  Month 3: number analyzed (Participants) | 220
  Month 3 | 55.9
  Month 6: number analyzed (Participants) | 192
  Month 6 | 69.3
  Month 12: number analyzed (Participants) | 156
  Month 12 | 66.0
  Month 18: number analyzed (Participants) | 135
  Month 18 | 71.9
  Month 24: number analyzed (Participants) | 118
  Month 24 | 73.7

6. Secondary Outcome: Percentage of Participants With LDA According to Simplified Disease Activity Index (SDAI) <=11
Description: SDAI is a composite end point, calculated as TJC + SJC (both using 28 joints) + PtGA (0-10 cm scale, higher score=more disease activity) + Physician Global Assessment (PhGA) (0-10 cm scale, higher score=more disease activity) + CRP (milligrams per deciliter [mg/dL]). The SDAI score is classified into four categories: remission (<=3.3), low (>3.3-11), moderate (>11-26), and high (>26) disease activity. The SDAI score ranges from 0 to 86 where higher scores indicates high disease activity. SDAI score of <=11 indicates LDA. Percentage of participants with SDAI <=11 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 272
  Baseline | 6.6
  Month 1: number analyzed (Participants) | 180
  Month 1 | 39.4
  Month 3: number analyzed (Participants) | 211
  Month 3 | 54.0
  Month 6: number analyzed (Participants) | 186
  Month 6 | 67.2
  Month 12: number analyzed (Participants) | 150
  Month 12 | 64.7
  Month 18: number analyzed (Participants) | 129
  Month 18 | 68.2
  Month 24: number analyzed (Participants) | 116
  Month 24 | 74.1

7. Secondary Outcome: Percentage of Participants With LDA According to Clinical Disease Activity Index (CDAI) <=10
Description: CDAI is a composite end point, calculated as TJC + SJC (both using 28 joints) + PtGA (0-10 cm scale, higher score=more disease activity) + PhGA (0-10 cm scale, higher score=more disease activity). The CDAI score is classified into four categories: remission (<=2.8), low (>2.8-10), moderate (>10-22), and high (>22) disease activity. The CDAI score ranges from 0 to 76, where higher scores indicates high disease activity. CDAI score of <=10 indicates LDA. Percentage of participants with CDAI <=10 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 280
  Baseline | 6.1
  Month 1: number analyzed (Participants) | 208
  Month 1 | 41.8
  Month 3: number analyzed (Participants) | 236
  Month 3 | 56.4
  Month 6: number analyzed (Participants) | 200
  Month 6 | 67.0
  Month 12: number analyzed (Participants) | 166
  Month 12 | 66.3
  Month 18: number analyzed (Participants) | 141
  Month 18 | 68.8
  Month 24: number analyzed (Participants) | 127
  Month 24 | 70.9

8. Secondary Outcome: Percentage of Participants With Remission According to DAS28-4 ESR<2.6
Description: DAS28-4 ESR is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (mm/h) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). The calculation of DAS28-4 ESR is as follows: 0.56 * sqrt (TJC) + 0.28 * sqrt (SJC) + 0.70* In(ESR) + 0.014* (PtGA); where ln = natural logarithm. Total DAS28-4 score range: 0 to 9.4, higher score=more disease activity. DAS28(ESR) score of <2.6 indicates LDA. Percentage of participants with DAS28-4 ESR <2.6 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 249
  Baseline | 3.6
  Month 1: number analyzed (Participants) | 152
  Month 1 | 17.8
  Month 3: number analyzed (Participants) | 196
  Month 3 | 27.6
  Month 6: number analyzed (Participants) | 166
  Month 6 | 34.9
  Month 12: number analyzed (Participants) | 135
  Month 12 | 32.6
  Month 18: number analyzed (Participants) | 116
  Month 18 | 33.6
  Month 24: number analyzed (Participants) | 103
  Month 24 | 38.8

9. Secondary Outcome: Percentage of Participants With Remission According to DAS28-4 CRP <2.6
Description: DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC with 28 joints assessed, SJC with 28 joints assessed, CRP (mg/L) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). The calculation of DAS28-4 CRP is as follows: 0.56 * sqrt (TJC) + 0.28 * sqrt (SJC) + 0.36 * ln (CRP+l) + 0.014*PtGA + 0.96; where ln = natural logarithm. Total DAS28-4 score range: 0 to 9.4, higher score=more disease activity. DAS28(CRP) score of <2.6 indicates LDA. Percentage of participants with DAS28-4 CRP <2.6 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 286
  Baseline | 4.9
  Month 1: number analyzed (Participants) | 184
  Month 1 | 29.3
  Month 3: number analyzed (Participants) | 220
  Month 3 | 37.3
  Month 6: number analyzed (Participants) | 192
  Month 6 | 46.4
  Month 12: number analyzed (Participants) | 156
  Month 12 | 48.1
  Month 18: number analyzed (Participants) | 135
  Month 18 | 48.9
  Month 24: number analyzed (Participants) | 118
  Month 24 | 59.3

10. Secondary Outcome: Percentage of Participants in Remission According to SDAI <=3.3
Description: SDAI is a composite end point, calculated as TJC + SJC (both using 28 joints) + PtGA (0-10 cm scale, higher score=more disease activity) + PhGA (0-10 cm scale, higher score=more disease activity) + CRP (mg/dL). The SDAI score is classified into four categories: remission (<=3.3), low (>3.3-11), moderate (>11-26), and high (>26) disease activity. The SDAI score ranges from 0 to 86 where higher scores indicates high disease activity. SDAI score of <=3.3 indicates LDA. Percentage of participants with SDAI <=3.3 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 272
  Baseline | 1.1
  Month 1: number analyzed (Participants) | 180
  Month 1 | 6.7
  Month 3: number analyzed (Participants) | 211
  Month 3 | 13.7
  Month 6: number analyzed (Participants) | 186
  Month 6 | 23.1
  Month 12: number analyzed (Participants) | 150
  Month 12 | 29.3
  Month 18: number analyzed (Participants) | 129
  Month 18 | 31.0
  Month 24: number analyzed (Participants) | 116
  Month 24 | 30.2

11. Secondary Outcome: Percentage of Participants in Remission According to CDAI<=2.8
Description: CDAI is a composite end point, calculated as TJC + SJC (both using 28 joints) + PtGA (0-10 cm scale) + PhGA (0-10 cm scale). The CDAI score is classified into four categories: remission (<=2.8), low (>2.8-10), moderate (>10-22), and high (>22) disease activity. The CDAI score ranges from 0 to 76, where higher scores indicates high disease activity. CDAI score of <=2.8 indicates LDA. Percentage of participants with CDAI <=2.8 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 280
  Baseline | 0.7
  Month 1: number analyzed (Participants) | 208
  Month 1 | 6.7
  Month 3: number analyzed (Participants) | 236
  Month 3 | 14.8
  Month 6: number analyzed (Participants) | 200
  Month 6 | 21.5
  Month 12: number analyzed (Participants) | 166
  Month 12 | 26.5
  Month 18: number analyzed (Participants) | 141
  Month 18 | 26.2
  Month 24: number analyzed (Participants) | 127
  Month 24 | 29.9

12. Secondary Outcome: Percentage of Participants With Remission According to American College of Rheumatology-European League Against Rheumatism (ACR-EULAR) 2011 Boolean Criteria
Description: ACREULAR 2011 Boolean criteria is derived as: ACR Remission = 1, if SJC (using 28 joints) <=1, TJC (using 28 joints) <=1, CRP <=1 mg/dL, and PtGA (0 to 10 cm scale, higher score=more disease activity) <=1 centimeter (cm) otherwise ACR remission =0. Higher scores indicated greater affection due to disease activity. Percentage of participants with remission according to ACR-EULAR 2011 Boolean criteria is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12 18, and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Percentage of participants
  Baseline: number analyzed (Participants) | 298
  Baseline | 2.7
  Month 1: number analyzed (Participants) | 190
  Month 1 | 8.9
  Month 3: number analyzed (Participants) | 228
  Month 3 | 14.9
  Month 6: number analyzed (Participants) | 205
  Month 6 | 22.0
  Month 12: number analyzed (Participants) | 167
  Month 12 | 24.6
  Month 18: number analyzed (Participants) | 143
  Month 18 | 26.6
  Month 24: number analyzed (Participants) | 123
  Month 24 | 24.4

13. Secondary Outcome: Change From Baseline in DAS28-4 ESR Score at Month 1, 3, 6, 12, 18 and 24
Description: DAS28-4 ESR is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (mm/h) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). The calculation of DAS28-4 ESR is as follows: 0.56 * sqrt (TJC) + 0.28 * sqrt (SJC) + 0.70* In(ESR) + 0.014* (PtGA); where ln = natural logarithm. Total DAS28-4 score range: 0 to 9.4, higher score=more disease activity. Mean change from baseline in DAS28-4 ESR score at months 3, 6, 12, 18 and 24 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 249
Units on a scale
  Baseline | 4.850 (1.180)
  Change at Month 1: number analyzed (Participants) | 135
  Change at Month 1 | -1.129 (1.187)
  Change at Month 3: number analyzed (Participants) | 170
  Change at Month 3 | -1.419 (1.487)
  Change at Month 6: number analyzed (Participants) | 150
  Change at Month 6 | -1.941 (1.367)
  Change at Month 12: number analyzed (Participants) | 119
  Change at Month 12 | -1.764 (1.347)
  Change at Month 18: number analyzed (Participants) | 99
  Change at Month 18 | -1.954 (1.487)
  Change at Month 24: number analyzed (Participants) | 85
  Change at Month 24 | -2.008 (1.363)

14. Secondary Outcome: Change From Baseline in DAS28-4 CRP Score at Month 1, 3, 6, 12, 18 and 24
Description: DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC with 28 joints assessed, SJC with 28 joints assessed, CRP (mg/L) and PtGA recorded on 100 mm VAS (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). The calculation of DAS28-4 CRP is as follows: 0.56 * sqrt (TJC) + 0.28 * sqrt (SJC) + 0.36 * ln (CRP+l) + 0.014*PtGA + 0.96; where ln = natural logarithm. Total DAS28-4 score range: 0 to 9.4, higher score=more disease activity. Mean change from baseline in DAS28-4 CRP score at months 3, 6, 12, 18 and 24 is presented in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 286
Units on a scale
  Baseline | 4.526 (1.088)
  Change at Month 1: number analyzed (Participants) | 177
  Change at Month 1 | -1.295 (1.135)
  Change at Month 3: number analyzed (Participants) | 211
  Change at Month 3 | -1.498 (1.363)
  Change at Month 6: number analyzed (Participants) | 185
  Change at Month 6 | -1.902 (1.198)
  Change at Month 12: number analyzed (Participants) | 148
  Change at Month 12 | -1.909 (1.269)
  Change at Month 18: number analyzed (Participants) | 125
  Change at Month 18 | -1.971 (1.275)
  Change at Month 24: number analyzed (Participants) | 111
  Change at Month 24 | -2.077 (1.215)

15. Secondary Outcome: Number of Participants Responding To Treatment by Considering DAS28 (EULAR Criterion)
Description: 28 EULAR criteria to evaluate participant's response to treatment is categorised as good responder, moderate responder and non-responder based on participants DAS28-4 CRP score and decrease in DAS28-4 CRP compared to initial pre-treatment visit (Visit 0 [V0]). Good response: DAS28 at treatment visit <= 3.2 and decrease in DAS 28 compared to V0 >1.2. Moderate responder: DAS28 at treatment visit > 3.2 to <= 5.1 or > 5.1 and decrease in DAS 28 compared to V0 >1.2 DAS28 at treatment visit <= 3.2 or > 3.2 to <= 5.1 and decrease in DAS 28 compared to V0 >0.6 and <=1.2. Non-responder: DAS28 at treatment visit > 5.1 and decrease in DAS 28 compared to V0 >0.6 to <=1.2 DAS28 at treatment visit <= 3.2 or > 3.2 to <= 5.1 or > 5.1 and decrease in DAS 28 compared to V0 <=0.6. Number of participants responding to treatment by considering DAS28 (EULAR criterion) is reported in this outcome measure.
Time Frame: Month 1, 3, 6, 12, 18, and 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Participants
  CRP, good responder, month 1: number analyzed (Participants) | 177
  CRP, good responder, month 1 | 67
  CRP, moderate responder, month 1: number analyzed (Participants) | 177
  CRP, moderate responder, month 1 | 61
  CRP, non-responder, month 1: number analyzed (Participants) | 177
  CRP, non-responder, month 1 | 49
  CRP, good responder, month 3: number analyzed (Participants) | 211
  CRP, good responder, month 3 | 97
  CRP, moderate responder, month 3: number analyzed (Participants) | 211
  CRP, moderate responder, month 3 | 63
  CRP, non-responder, month 3: number analyzed (Participants) | 211
  CRP, non-responder, month 3 | 51
  CRP, good responder, month 6: number analyzed (Participants) | 185
  CRP, good responder, month 6 | 111
  CRP, moderate responder, month 6: number analyzed (Participants) | 185
  CRP, moderate responder, month 6 | 47
  CRP, non-responder, month 6: number analyzed (Participants) | 185
  CRP, non-responder, month 6 | 27
  CRP, good responder, month 12: number analyzed (Participants) | 148
  CRP, good responder, month 12 | 84
  CRP, moderate responder, month 12: number analyzed (Participants) | 148
  CRP, moderate responder, month 12 | 41
  CRP, non-responder, month 12: number analyzed (Participants) | 148
  CRP, non-responder, month 12 | 23
  CRP, good responder, month 18: number analyzed (Participants) | 125
  CRP, good responder, month 18 | 78
  CRP, moderate responder, month 18: number analyzed (Participants) | 125
  CRP, moderate responder, month 18 | 24
  CRP, non-responder, month 18: number analyzed (Participants) | 125
  CRP, non-responder, month 18 | 23
  CRP, good responder, month 24: number analyzed (Participants) | 111
  CRP, good responder, month 24 | 70
  CRP, moderate responder, month 24: number analyzed (Participants) | 111
  CRP, moderate responder, month 24 | 28
  CRP, non-responder, month 24: number analyzed (Participants) | 111
  CRP, non-responder, month 24 | 13
  ESR, good responder, month 1: number analyzed (Participants) | 135
  ESR, good responder, month 1 | 37
  ESR, moderate responder, month 1: number analyzed (Participants) | 135
  ESR, moderate responder, month 1 | 50
  ESR, non-responder, month 1: number analyzed (Participants) | 135
  ESR, non-responder, month 1 | 48
  ESR, good responder, month 3: number analyzed (Participants) | 170
  ESR, good responder, month 3 | 59
  ESR, moderate responder, month 3: number analyzed (Participants) | 170
  ESR, moderate responder, month 3 | 56
  ESR, non-responder, month 3: number analyzed (Participants) | 170
  ESR, non-responder, month 3 | 55
  ESR, good responder, month 6: number analyzed (Participants) | 150
  ESR, good responder, month 6 | 65
  ESR, moderate responder, month 6: number analyzed (Participants) | 150
  ESR, moderate responder, month 6 | 62
  ESR, non-responder, month 6: number analyzed (Participants) | 150
  ESR, non-responder, month 6 | 23
  ESR, good responder, month 12: number analyzed (Participants) | 119
  ESR, good responder, month 12 | 55
  ESR, moderate responder, month 12: number analyzed (Participants) | 119
  ESR, moderate responder, month 12 | 40
  ESR, non-responder, month 12: number analyzed (Participants) | 119
  ESR, non-responder, month 12 | 24
  ESR, good responder, month 18: number analyzed (Participants) | 99
  ESR, good responder, month 18 | 51
  ESR, moderate responder, month 18: number analyzed (Participants) | 99
  ESR, moderate responder, month 18 | 30
  ESR, non-responder, month 18: number analyzed (Participants) | 99
  ESR, non-responder, month 18 | 18
  ESR, good responder, month 24: number analyzed (Participants) | 85
  ESR, good responder, month 24 | 43
  ESR, moderate responder, month 24: number analyzed (Participants) | 85
  ESR, moderate responder, month 24 | 28
  ESR, non-responder, month 24: number analyzed (Participants) | 85
  ESR, non-responder, month 24 | 14

16. Secondary Outcome: Change From Baseline in TJC at Month 1, 3, 6, 12, 18 and 24
Description: TJC (28) is the count of the total number of tender joints out of a possible 28 joints which are checked at the visit. TJC was used to measure the pain and inflammation in the joints. Mean change from baseline in TJC is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | Tofacitinib
Number analyzed (Participants) | 302
Tender Joints
  Baseline | 7.4 (6.0)
  Change at Month 1: number analyzed (Participants) | 213
  Change at Month 1 | -4.2 (5.8)
  Change at Month 3: number analyzed (Participants) | 245
  Change at Month 3 | -4.3 (6.5)
  Change at Month 6: number analyzed (Participants) | 214
  Change at Month 6 | -4.9 (6.3)
  Change at Month 12: number analyzed (Participants) | 175
  Change at Month 12 | -5.0 (7.0)
  Change at Month 18: number analyzed (Participants) | 153
  Change at Month 18 | -5.1 (5.9)
  Change at Month 24: number analyzed (Participants) | 131
  Change at Month 24 | -5.1 (6.7)

17. Secondary Outcome: Change From Baseline in SJC at Month 1, 3, 6, 12, 18 and 24
Description: SJC (28) is the count of the total number of swollen joints out of a possible 28 joints which are checked at the visit. SJC was used to measure the pain and inflammation in the joints. Mean change from baseline in TJC is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | Tofacitinib
Number analyzed (Participants) | 302
Swollen Joints
  Baseline | 5.3 (5.1)
  Change at Month 1: number analyzed (Participants) | 214
  Change at Month 1 | -3.0 (4.5)
  Change at Month 3: number analyzed (Participants) | 245
  Change at Month 3 | -3.5 (4.9)
  Change at Month 6: number analyzed (Participants) | 212
  Change at Month 6 | -3.9 (5.1)
  Change at Month 12: number analyzed (Participants) | 175
  Change at Month 12 | -4.3 (5.1)
  Change at Month 18: number analyzed (Participants) | 153
  Change at Month 18 | -4.4 (5.2)
  Change at Month 24: number analyzed (Participants) | 131
  Change at Month 24 | -4.3 (5.1)

18. Secondary Outcome: Number of Participants With Fibromyalgia Rapid Screening Tool (FiRST) Questionnaire Response
Description: FiRST is used to detect fibromyalgia in participants with diffuse rheumatic pain. It is a questionnaire which contains 6 items: diffuse pain, painful symptoms, fatigue, sleep and cognitive disorders, nonpainful abnormal sensations and functional somatic symptoms. Each of the 6 items contain yes or no response, and a positive answer to 5 out of the 6 answers can detect fibromyalgia. At each specified time points number of participants with "Yes" or "No" to fibromyalgia is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18 and 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Participants
  Baseline, Fibromyalgia: No: number analyzed (Participants) | 247
  Baseline, Fibromyalgia: No | 156
  Baseline, Fibromyalgia: Yes: number analyzed (Participants) | 247
  Baseline, Fibromyalgia: Yes | 91
  Month 1, Fibromyalgia: No: number analyzed (Participants) | 184
  Month 1, Fibromyalgia: No | 124
  Month 1, Fibromyalgia: Yes: number analyzed (Participants) | 184
  Month 1, Fibromyalgia: Yes | 60
  Month 3, Fibromyalgia: No: number analyzed (Participants) | 205
  Month 3, Fibromyalgia: No | 149
  Month 3, Fibromyalgia: Yes: number analyzed (Participants) | 205
  Month 3, Fibromyalgia: Yes | 56
  Month 6, Fibromyalgia: No: number analyzed (Participants) | 176
  Month 6, Fibromyalgia: No | 135
  Month 6, Fibromyalgia: Yes: number analyzed (Participants) | 176
  Month 6, Fibromyalgia: Yes | 41
  Month 12, Fibromyalgia: No: number analyzed (Participants) | 143
  Month 12, Fibromyalgia: No | 111
  Month 12, Fibromyalgia: Yes: number analyzed (Participants) | 143
  Month 12, Fibromyalgia: Yes | 32
  Month 18, Fibromyalgia: No: number analyzed (Participants) | 114
  Month 18, Fibromyalgia: No | 89
  Month 18, Fibromyalgia: Yes: number analyzed (Participants) | 114
  Month 18, Fibromyalgia: Yes | 25
  Month 24, Fibromyalgia: No: number analyzed (Participants) | 105
  Month 24, Fibromyalgia: No | 80
  Month 24, Fibromyalgia: Yes: number analyzed (Participants) | 105
  Month 24, Fibromyalgia: Yes | 25

19. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Month 1, 3, 6, 12, 18 and 24
Description: Morning stiffness is a common symptom of rheumatoid arthritis. The duration of morning stiffness is measured in minutes. Mean change from baseline in morning stiffness is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tofacitinib
Number analyzed (Participants) | 287
Minutes
  Baseline | 51.5 (53.3)
  Change at Month 1: number analyzed (Participants) | 202
  Change at Month 1 | -24.3 (43.0)
  Change at Month 3: number analyzed (Participants) | 234
  Change at Month 3 | -31.3 (48.8)
  Change at Month 6: number analyzed (Participants) | 198
  Change at Month 6 | -31.5 (49.1)
  Change at Month 12: number analyzed (Participants) | 163
  Change at Month 12 | -36.6 (50.8)
  Change at Month 18: number analyzed (Participants) | 130
  Change at Month 18 | -32.2 (47.9)
  Change at Month 24: number analyzed (Participants) | 117
  Change at Month 24 | -40.0 (49.3)

20. Secondary Outcome: Number of Participants Based on Response to Girerd Questionnaire at Month 1, 3, 6, 12, 18 and 24
Description: Girerd questionnaire is used to evaluate participant's treatment compliance and is made up of 6 yes or no questions. lf the participant responds "no" to all questions, it is considered as participant is a good complier. lf the participant responds "yes" once or twice, it is considered as participant is a minor complier. lf the participant responds "yes" three times or more, it is considered as participant is a no-complier.
Time Frame: Month 1, 3, 6, 12, 18 and 24
Population: Full analysis set population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Participants
  Good complier at baseline: number analyzed (Participants) | 256
  Good complier at baseline | 100
  Minor complier at baseline: number analyzed (Participants) | 256
  Minor complier at baseline | 139
  No-complier at baseline: number analyzed (Participants) | 256
  No-complier at baseline | 17
  Good complier at month 1: number analyzed (Participants) | 187
  Good complier at month 1 | 89
  Minor complier at month 1: number analyzed (Participants) | 187
  Minor complier at month 1 | 91
  No-complier at month 1: number analyzed (Participants) | 187
  No-complier at month 1 | 7
  Good complier at month 3: number analyzed (Participants) | 211
  Good complier at month 3 | 87
  Minor complier at month 3: number analyzed (Participants) | 211
  Minor complier at month 3 | 110
  No-complier at month 3: number analyzed (Participants) | 211
  No-complier at month 3 | 14
  Good complier at month 6: number analyzed (Participants) | 182
  Good complier at month 6 | 58
  Minor complier at month 6: number analyzed (Participants) | 182
  Minor complier at month 6 | 106
  No-complier at month 6: number analyzed (Participants) | 182
  No-complier at month 6 | 18
  Good complier at month 12: number analyzed (Participants) | 149
  Good complier at month 12 | 58
  Minor complier at month 12: number analyzed (Participants) | 149
  Minor complier at month 12 | 85
  No-complier at month 12: number analyzed (Participants) | 149
  No-complier at month 12 | 6
  Good complier at month 18: number analyzed (Participants) | 121
  Good complier at month 18 | 49
  Minor complier at month 18: number analyzed (Participants) | 121
  Minor complier at month 18 | 63
  No-complier at month 18: number analyzed (Participants) | 121
  No-complier at month 18 | 9
  Good complier at month 24: number analyzed (Participants) | 109
  Good complier at month 24 | 42
  Minor complier at month 24: number analyzed (Participants) | 109
  Minor complier at month 24 | 62
  No-complier at month 24: number analyzed (Participants) | 109
  No-complier at month 24 | 5

21. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQoL) 5-Dimension 3 Levels of Severity (EQ-5D-3L) Index Score at Month 1, 3, 6, 12, 18 and 24
Description: EQ-5D-3L is a standardized, participant administered measure of self-reported instrument used to evaluate health-related quality of life. It consists of two parts: EQ-5D index score (Part I) and the EQ-VAS (Part II). For Part I, i.e. EQ-5D-3L index score, participants rated their current health state on 5 single-item dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with each dimension having three levels of function:. 1=no problems, 2=some problems and 3=extreme problems. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score was transformed and results in a total index score range of 0 to 1.00; higher scores indicating a better health condition. Mean change from baseline in EQ-5D-3L index score is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 257
Units on a scale
  Baseline | 0.3987 (0.3731)
  Change at Month 1: number analyzed (Participants) | 179
  Change at Month 1 | 0.1314 (0.3185)
  Change at Month 3: number analyzed (Participants) | 203
  Change at Month 3 | 0.1767 (0.4054)
  Change at Month 6: number analyzed (Participants) | 176
  Change at Month 6 | 0.1886 (0.3638)
  Change at Month 12: number analyzed (Participants) | 142
  Change at Month 12 | 0.2362 (0.4058)
  Change at Month 18: number analyzed (Participants) | 119
  Change at Month 18 | 0.2190 (0.4020)
  Change at Month 24: number analyzed (Participants) | 106
  Change at Month 24 | 0.2123 (0.3911)

22. Secondary Outcome: Change From Baseline in Short Form-12 Health Survey (SF-12) Score at Month 1, 3, 6, 12, 18 and 24
Description: SF-12 was a participant reported outcome survey that represented overall health status by measuring 8 health-related aspects of an individual: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE) and Mental Health (MH). The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Responses on the SF-12 were also used to calculate 2 summary scores: Physical component score (PCS) and mental component score (MCS). The score range for each of these 2 summary scores was from 0 (poor health) to 100 (better health), where 100 indicated good health condition. Mean change from baseline in PCS and MCS scores are reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18 and 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 306
Units on a scale
  PCS at Baseline: number analyzed (Participants) | 246
  PCS at Baseline | 35.0 (8.7)
  PCS at Change at Month 1: number analyzed (Participants) | 166
  PCS at Change at Month 1 | 3.5 (7.6)
  PCS at Change at Month 3: number analyzed (Participants) | 186
  PCS at Change at Month 3 | 5.8 (8.9)
  PCS at Change at Month 6: number analyzed (Participants) | 164
  PCS at Change at Month 6 | 5.9 (8.7)
  PCS at Change at Month 12: number analyzed (Participants) | 130
  PCS at Change at Month 12 | 6.9 (9.2)
  PCS at Change at Month 18: number analyzed (Participants) | 113
  PCS at Change at Month 18 | 6.9 (9.1)
  PCS at Change at Month 24: number analyzed (Participants) | 100
  PCS at Change at Month 24 | 7.3 (9.8)
  MCS at Baseline: number analyzed (Participants) | 246
  MCS at Baseline | 40.2 (10.4)
  MCS at Change at Month 1: number analyzed (Participants) | 166
  MCS at Change at Month 1 | 1.7 (9.1)
  MCS at Change at Month 3: number analyzed (Participants) | 186
  MCS at Change at Month 3 | 3.7 (10.6)
  MCS at Change at Month 6: number analyzed (Participants) | 164
  MCS at Change at Month 6 | 3.9 (9.5)
  MCS at Change at Month 12: number analyzed (Participants) | 130
  MCS at Change at Month 12 | 3.9 (11.1)
  MCS at Change at Month 18: number analyzed (Participants) | 113
  MCS at Change at Month 18 | 4.0 (10.2)
  MCS at Change at Month 24: number analyzed (Participants) | 100
  MCS at Change at Month 24 | 4.9 (10.7)

23. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Total Score at Month 1, 3, 6, 12, 18 and 24
Description: FACIT-Fatigue questionnaire consists of 13 self-evaluated questions. Each question has a response of values 0 (not at all) to 4 (very much). Score for each question is calculated by first reversing negatively stated-items (subtracting the response from '4' except for the 2 positively stated-items) and then summing the raw (0-4) scores. The FACIT-Fatigue total score is derived by summing the response to each question which gives a value between 0 (worse score) and 52 (best score). Higher scores represent better participant's status (less fatigue). Mean change from baseline in FACIT-Fatigue total score is reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 18 and 24
Population: Full analysis set population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. Here, "Number of participants analyzed" signifies number of participants evaluable and contributed to data for this outcome measure. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 259
Units on a scale
  Baseline | 26.9 (11.7)
  Change at Month 1: number analyzed (Participants) | 183
  Change at Month 1 | 3.9 (9.3)
  Change at Month 3: number analyzed (Participants) | 205
  Change at Month 3 | 6.2 (10.9)
  Change at Month 6: number analyzed (Participants) | 179
  Change at Month 6 | 6.2 (10.1)
  Change at Month 12: number analyzed (Participants) | 145
  Change at Month 12 | 6.9 (12.1)
  Change at Month 18: number analyzed (Participants) | 121
  Change at Month 18 | 6.8 (11.6)
  Change at Month 24: number analyzed (Participants) | 107
  Change at Month 24 | 8.4 (11.4)

24. Secondary Outcome: Number of Participants With Tofacitinib Tolerance Issue
Description: Number of participants who discontinued tofacitinib due to tolerance issue.
Time Frame: Month 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 309
Participants | 39

ADVERSE EVENTS:
Time Frame: Baseline up to 24 months after Tofacitinib treatment initiation (for a maximum of 48 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 3/309
Serious Adverse Events (participants affected / at risk) | 64/309
Other Adverse Events (participants affected / at risk) | 197/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=309)
ANAEMIA (Blood and lymphatic system disorders) | 1
LYMPHOPROLIFERATIVE DISORDER (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
PERICARDITIS (Cardiac disorders) | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 1
DEATH (General disorders) | 1
DRUG INEFFECTIVE (General disorders) | 1
DRUG THERAPEUTIC INCOMPATIBILITY (General disorders) | 1
INFLAMMATION (General disorders) | 1
MALAISE (General disorders) | 1
TREATMENT FAILURE (General disorders) | 1
TUMOUR OF AMPULLA OF VATER (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 3
APPENDICITIS (Infections and infestations) | 2
ABSCESS (Infections and infestations) | 1
ABSCESS LIMB (Infections and infestations) | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 1
CAMPYLOBACTER SEPSIS (Infections and infestations) | 1
ENDOCARDITIS (Infections and infestations) | 1
HELICOBACTER INFECTION (Infections and infestations) | 1
HEPATITIS E (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 1
LATENT TUBERCULOSIS (Infections and infestations) | 1
PAROTITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
TUBERCULOSIS (Infections and infestations) | 1
SHOULDER FRACTURE (Injury, poisoning and procedural complications) | 2
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1
MEDICATION ERROR (Injury, poisoning and procedural complications) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 1
PLATELET COUNT DECREASED (Investigations) | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SMALL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2
INTRACRANIAL MASS (Nervous system disorders) | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1
PREGNANCY, PUERPERIUM AND PERINATAL CONDITIONS (Pregnancy, puerperium and perinatal conditions) | 1
COMPLETED SUICIDE (Psychiatric disorders) | 1
NEPHROPATHY TOXIC (Renal and urinary disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
MITRAL VALVE REPLACEMENT (Surgical and medical procedures) | 1
SPINAL FUSION SURGERY (Surgical and medical procedures) | 1
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=309)
LYMPHOPENIA (Blood and lymphatic system disorders) | 4
ANAEMIA (Blood and lymphatic system disorders) | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 3
PALPITATIONS (Cardiac disorders) | 4
TACHYCARDIA (Cardiac disorders) | 2
VERTIGO (Ear and labyrinth disorders) | 4
TINNITUS (Ear and labyrinth disorders) | 1
THYROID MASS (Endocrine disorders) | 1
GLARE (Eye disorders) | 1
NAUSEA (Gastrointestinal disorders) | 11
VOMITING (Gastrointestinal disorders) | 7
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
DYSPEPSIA (Gastrointestinal disorders) | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
APHTHOUS ULCER (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
EPIPLOIC APPENDAGITIS (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
HIATUS HERNIA (Gastrointestinal disorders) | 1
TREATMENT FAILURE (General disorders) | 44
DRUG INEFFECTIVE (General disorders) | 12
ASTHENIA (General disorders) | 5
FATIGUE (General disorders) | 5
OEDEMA PERIPHERAL (General disorders) | 4
CHEST DISCOMFORT (General disorders) | 3
CHEST PAIN (General disorders) | 3
PYREXIA (General disorders) | 2
THERAPEUTIC RESPONSE SHORTENED (General disorders) | 2
DRUG INTOLERANCE (General disorders) | 1
FACE OEDEMA (General disorders) | 1
FEELING DRUNK (General disorders) | 1
FEELING OF BODY TEMPERATURE CHANGE (General disorders) | 1
INFLAMMATION (General disorders) | 1
INFLUENZA LIKE ILLNESS (General disorders) | 1
INJECTION SITE PAIN (General disorders) | 1
MALAISE (General disorders) | 1
PAIN (General disorders) | 1
SWELLING FACE (General disorders) | 1
HEPATIC CYTOLYSIS (Hepatobiliary disorders) | 4
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 4
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1
BRONCHITIS (Infections and infestations) | 15
HERPES ZOSTER (Infections and infestations) | 13
URINARY TRACT INFECTION (Infections and infestations) | 8
NASOPHARYNGITIS (Infections and infestations) | 6
INFLUENZA (Infections and infestations) | 5
SINUSITIS (Infections and infestations) | 5
TOOTH INFECTION (Infections and infestations) | 3
GINGIVITIS (Infections and infestations) | 2
HORDEOLUM (Infections and infestations) | 2
ORAL HERPES (Infections and infestations) | 2
PARONYCHIA (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 2
TOOTH ABSCESS (Infections and infestations) | 2
ARTHRITIS INFECTIVE (Infections and infestations) | 1
CHRONIC SINUSITIS (Infections and infestations) | 1
CONJUNCTIVITIS (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 1
DERMATITIS INFECTED (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
GENITAL HERPES (Infections and infestations) | 1
GENITAL INFECTION FUNGAL (Infections and infestations) | 1
HERPES DERMATITIS (Infections and infestations) | 1
HERPES VIRUS INFECTION (Infections and infestations) | 1
LARYNGITIS (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
RECTAL ABSCESS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 1
RHINOTRACHEITIS (Infections and infestations) | 1
SINUSITIS BACTERIAL (Infections and infestations) | 1
SKIN INFECTION (Infections and infestations) | 1
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1
TINEA MANUUM (Infections and infestations) | 1
TONSILLITIS (Infections and infestations) | 1
TRACHEITIS (Infections and infestations) | 1
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 2
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1
BURN ORAL CAVITY (Injury, poisoning and procedural complications) | 1
BURSITIS (Injury, poisoning and procedural complications) | 1
EYELID INJURY (Injury, poisoning and procedural complications) | 1
PRODUCT DOSE OMISSION IN ERROR (Injury, poisoning and procedural complications) | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1
WEIGHT INCREASED (Investigations) | 5
LABORATORY TEST ABNORMAL (Investigations) | 2
TRANSAMINASES INCREASED (Investigations) | 2
BLOOD PRESSURE ABNORMAL (Investigations) | 1
BLOOD UREA INCREASED (Investigations) | 1
CORONAVIRUS TEST POSITIVE (Investigations) | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 1
PREGNANCY TEST POSITIVE (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 4
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
BURSITIS (Musculoskeletal and connective tissue disorders) | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 2
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HEADACHE (Nervous system disorders) | 14
SCIATICA (Nervous system disorders) | 3
MIGRAINE (Nervous system disorders) | 2
NEURALGIA (Nervous system disorders) | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1
NIGHTMARE (Psychiatric disorders) | 1
GLOMERULONEPHRITIS MEMBRANOUS (Renal and urinary disorders) | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 4
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 4
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1
LUNG OPACITY (Respiratory, thoracic and mediastinal disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 6
ALOPECIA (Skin and subcutaneous tissue disorders) | 2
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 2
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 2
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 1
PRURIGO (Skin and subcutaneous tissue disorders) | 1
SKIN BURNING SENSATION (Skin and subcutaneous tissue disorders) | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1
DENTAL IMPLANTATION (Surgical and medical procedures) | 1
THERAPY CESSATION (Surgical and medical procedures) | 1
FLUSHING (Vascular disorders) | 1
HAEMATOMA (Vascular disorders) | 1
HOT FLUSH (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 1
PHLEBITIS (Vascular disorders) | 1
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT03981900/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03981900/SAP_001.pdf